CLINICAL TRIAL: NCT07339566
Title: Efficacy and Safety of Xeligekimab in the Treatment of Non-Radiographic Axial Spondyloarthritis: A Single-Center, Single-Arm Study
Brief Title: Efficacy and Safety of Xeligekimab in the Treatment of Non-Radiographic Axial Spondyloarthritis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lingli Dong (Other)
Responsible Party: Sponsor-Investigator, Lingli Dong, professor;professor of medicine, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nr-axSpA--IL17Ai
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nr-axial Spondyloarthritis; Non-Radiographical Axial Spondyloarthritis
Keywords: Nr-axSpA; Xeligekimab Injection; IL-17A
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xeligekimab treatment (Experimental): Through the subcutaneous administration of Xeligekimab, it is hoped to achieve the control of symptoms and inflammation in nr-axSpA, prevent or delay structural damage, and maximize patients' quality of life.
  Interventions: Drug: Xeligekimab injection

INTERVENTIONS:
Drug: Xeligekimab injection — Subjects who have signed the informed consent form will undergo examinations and assessments according to the inclusion/exclusion criteria specified in the trial protocol. After screening and successful enrollment, they will enter the treatment period. Dosing time points are (W0, W2, W4, W8, W12), with a subcutaneous injection of Xeligekimab 100mg each time. Week 12 is the last dosing time. After week 12, the physician will comprehensively assess whether to continue using Xeligekimab based on the patient's condition. If continuation is required, the patient will need to purchase Xeligekimab at their own expense.
  During the trial, the research physician and nurse will monitor safety, record the subject's vital signs and adverse events after dosing. Laboratory tests will be performed before and after the trial.

SUMMARY:
Subjects who have signed the informed consent form will undergo examinations and assessments according to the inclusion/exclusion criteria specified in the trial protocol. After screening and successful enrollment, they will enter the treatment period. Dosing time points are (W0, W2, W4, W8, W12), with a subcutaneous injection of Xeligekimab 100mg each time. Week 12 is the last dosing time. After week 12, the physician will comprehensively assess whether to continue using Xeligekimab based on the patient's condition. If continuation is required, the patient will need to purchase Xeligekimab at their own expense.

During the trial, the research physician and nurse will monitor safety, record the subject's vital signs and adverse events after dosing. Laboratory tests will be performed before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older;
* Diagnosis of non-radiographic axial spondyloarthritis (nr-axSpA) according to the Assessment of SpondyloArthritis International Society (ASAS) criteria for axial spondyloarthritis;
* Ineffective or intolerant to NSAID therapy;
* Objective signs of inflammation (abnormal MRI or C-reactive protein);
* Active axial spondyloarthritis with BASDAI score ≥4 and BASDAI question 2 ≥4;
* Visual Analogue Scale (VAS) score ≥4;

Exclusion Criteria:

* Patients with radiographic evidence of sacroiliitis, bilateral ≥grade 2 or unilateral ≥grade 3;
* Presence of other active inflammations besides axial spondyloarthritis (e.g., active inflammatory bowel disease [IBD] or uveitis);
* Chest X-ray suggesting active infection or malignant lesions;
* Active systemic infection within 2 weeks prior to enrollment;
* Known tuberculosis, HIV, hepatitis B, or hepatitis C infection at screening;
* History of lymphoproliferative disease, any history of malignancy (within the past 5 years);
* Subjects with unstable cardiovascular disease;
* Patients taking potent opioid analgesics;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving ASAS20 (ankylosing spondylitis disease activity score) at week 12 | at the 12th week after administration
  ASAS20 response is defined as an improvement of
  20% and an absolute improvement from baseline of 2 units on a 10-point scale in at least three of the four main domains and no worsening assessed at all in the remaining domain.
  Main ASAS domains:
  Patient's global assessment of disease activity measured on a VAS scale Patient's assessment of back pain, represented by either total or nocturnal pain scores, both measured on a VAS scale Function represented by BASFI average of 10 questions regarding ability to perform specific tasks as measured by VAS scale Inflammation represented by mean duration and severity of morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI as measured by VAS scale

SECONDARY OUTCOMES:
The proportion of overall participants achieving an ASAS40 response at week 12. | week 12
  ASAS40 response is defined as an improvement of
  40% and an absolute improvement from baseline of 2 units on a 10-point scale in at least three of the four main domains and no worsening assessed at all in the remaining domain.
The proportion of participants meeting the ASAS 5/6 response criteria. | week 12
  ASAS 5/6 response is defined as an improvement of
  ≥20% in at least five of all six domains.
The change from baseline in total Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). | week 12
  The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) consists of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which is used to answer 6 questions pertaining to the 5 major symptoms of AS.
The change from baseline in total Bath Ankylosing Spondylitis Functional Index (BASFI). | week 12
  The BASFI (Bath Ankylosing Spondylitis Functional Index) is a set of 10 questions designed to determine the degree of functional limitation in those patients with AS.
The change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL) scores. | week 12
  The ASQoL (Ankylosing Spondylitis Quality of Life scores) is an instrument to measure health-related quality of life among patients with Ankylosig spondylosrthritis.
Incidents of AE、TRAE、SAE | up to 12 weeks
  overall safety and tolerability of Xeligekimab.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No